CLINICAL TRIAL: NCT05543018
Title: Effect of Intraocular Tamponade on Visual Function in the Human Eyes
Brief Title: Effect of Intraocular Tamponade on Visual Perception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-10-22
Record Dates: First submitted 2022-09-12; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Retinal Detachment; Optic Neuropathy; Glaucoma
Keywords: Vitrectomy; Retinal detachment; Intraocular Tamponade; Silicon oil; Air tamponade
MeSH Terms: conditions — Retinal Detachment; Optic Nerve Diseases; Glaucoma | interventions — Electroretinography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silicon oil group (Active Comparator): Patients diagnosed with retinal detachment and undergone vitrectomy operation with silicon oil tamponade.
  Interventions: Diagnostic Test: Electroretinogram; Procedure: Vitrectomy operation
- Air tamponade (Active Comparator): Patients diagnosed with retinal detachment and undergone vitrectomy operation with air tamponade.
  Interventions: Diagnostic Test: Electroretinogram; Procedure: Vitrectomy operation
- Non-expansile gas (Active Comparator): Patients diagnosed with retinal detachment and undergone vitrectomy operation with non-expansile gas tamponade (sulfur hexafluoride).
  Interventions: Diagnostic Test: Electroretinogram; Procedure: Vitrectomy operation

INTERVENTIONS:
Diagnostic Test: Electroretinogram — Retinal function assessment using electroretinogram
Procedure: Vitrectomy operation — Vitrectomy operation to treat retinal detachment

SUMMARY:
Intraocular tamponade used in vitrectomy operations may affects retinal function in various mechanisms.

DETAILED DESCRIPTION:
Various intraocular tamponade are being used in vitrectomy operations as gases, fluids and silicon oil. The effects of these intraocular tamponade may affects the final visual outcome of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* primary retinal detachment patients.
* patients eligible for 23 gauge pars-plana vitrectomy operation.

Exclusion Criteria:

* patients with axial length more than 30 millimeter that may have severe chorioretinal degenerations that may affects retinal function.
* patients with macular diseases that may affects final visual outcome as macular holes and choroidal neovascular membranes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-28 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Baseline and monthly after surgery till 6 months of follow up.
  Changes in visual acuity measured in LogMAR units.
Retinal function amplitude | Baseline and monthly after surgery till 6 months of follow up.
  Changes in electroretinogram amplitude parameters in microvolt/second measured by roland consult retinal function device.
Retinal function implicit time. | Baseline and monthly after surgery till 6 months of follow up.
  Changes in electroretinogram implicit time in millisecond measured by roland consult retinal function device.

SECONDARY OUTCOMES:
Intraocular pressure | Baseline and monthly after surgery till 6 months of follow up.
  Changes in intraocular pressure measured by goldman applanation tonometry in millimeter mercury.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: No